CLINICAL TRIAL: NCT01141530
Title: Deep Sequencing of the Breast Cancer Transcriptome
Status: Withdrawn | Type: Observational
Why Stopped: Study withdrawn due to inability to enroll subjects.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 111481
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Breast Cancer
Keywords: Identify novel genes and predict putative proteins in breast cancer.; Find biomarkers that can be used for early detection, diagnosis, and prognosis.
MeSH Terms: conditions — Breast Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The informed consent process for biospecimen collection we expect to use in this research has already been obtained by the UAMS Tissue Bank personnel as a part of the UARK 2005-06 protocol. Tissue is collected during biopsies or mastectomies after pathologist approval. We will sequence small non-coding molecules (microRNA), messenger RNA, chromatin immunoprecipated and bisulfite treated DNA.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Tissue Bank Samples: Because this study is a retrospective tissue bank study, there are no subjects actively participating in this study. All samples studied will be obtained through the UAMS Tissue Bank.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Because this study is a retrospective tissue bank study, there are no subjects actively participating in this study, thus no intervention. All samples studied will be obtained through the UAMS Tissue Bank.

SUMMARY:
This project is a pilot study designed to investigate transcriptional regulation in breast cancer. Although the main focus of the present study will be triple negative breast cancer where all of the clinically relevant receptors - estrogen receptor (ER), progesterone receptor (PR) and herceptin (HER2) - are absent, all breast tissue biospecimens, including normal and mammary dysplasia, stored in the UAMS Tissue bank, procured from outside collaborators or purchased from commercial vendors will eventually be investigated. We will use high throughput molecular profiling techniques such as microarrays and next generation sequencing to correlate gene expression and gene expression regulation with clinical parameters such as tumor size, time to relapse and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* There is no inclusion criteria. This study is a retrospective tissue bank study analyzing tissue collected from a previous clinical trial. No subjects will be enrolled.

Exclusion Criteria:

* There is no exclusion criteria. This study is a retrospective tissue bank study analyzing tissue collected from a previous clinical trial. No subjects will be enrolled.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a retrospective tissue bank study analyzing tissue collected from a previous clinical trial. No subjects will be enrolled. Tissue was collected during biopsies or mastectomies after pathologist's approval.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States